CLINICAL TRIAL: NCT03814577
Title: A Comparison of the Effects of Desflurane and Total Intravenous Anesthesia (TIVA) on Antioxidant System in Morbidly Obese Patients Undergoing Bariatric Surgery: A Randomized Trial
Brief Title: A Comparison of the Effects of Desflurane and TIVA on Antioxidant System in Morbidly Obese Patients
Acronym: OxSys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sedat AKBAS, Asst. Prof. Dr. Sedat Akbas, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: sedatakbas6
Record Dates: First submitted 2019-01-07; First posted 2019-01-24 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Oxidative Stress; Morbid Obesity
Keywords: General anesthesia; Inhalation anesthetics; Total Intravenous anesthesia; Oxidative Stress; Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Consciousness Monitors

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Clinical Study
Masking Description: Single (Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desflurane (Active Comparator): Anesthesia will be maintained with Desflurane inhalation with a flow of 2 L/min in 0.5 O2 oxygen air mixture.Total Intravenous Anesthesia will not be used in this group. While target desflurane minimum alveolar concentration (MAC) will be 1-1.5 and Bispectral Index values will be between 40-60, the flow rate will be adjusted to 2 L/min. Total Antioxidant Status and Total Oxidant Status will be then measured. Invasive arterial monitorization will be performed to right radial artery under local anesthesia to follow up hemodynamic changes and take the blood samples.
  Interventions: Diagnostic Test: Total Antioxidant Status; Diagnostic Test: Total Oxidant Status; Device: Bispectral Index; Other: Invasive arterial monitorization
- Total Intravenous Anesthesia (Experimental): Total Intravenous Anesthesia: Anesthesia will be maintained with inhalation with a flow of 2 L/min in 0.5 O2 oxygen air mixture. Desflurane will not be used in this group. Total Intravenous Anesthesia (propofol and remifentanyl infusion) will be performed to the patients while target Bispectral Index values were between 40-60. Also the flow rate will be adjusted to 2 L/min. Total Antioxidant Status and Total Oxidant Status will be then measured. Invasive arterial monitorization will be performed to right radial artery under local anesthesia to follow up hemodynamic changes and take the blood samples.
  Interventions: Diagnostic Test: Total Antioxidant Status; Diagnostic Test: Total Oxidant Status; Device: Bispectral Index; Other: Invasive arterial monitorization

INTERVENTIONS:
Diagnostic Test: Total Antioxidant Status — Total Antioxidant Status values will be determined using a novel automated measurement method. The colour intensity, which can be measured spectrophotometrically, is related to the total amount of oxidant molecules present in the sample. The assay is calibrated with hydrogen peroxide) and the results are expressed in terms of micromolar hydrogen peroxide equivalent per litre.
Diagnostic Test: Total Oxidant Status — Total Oxidant Status values will be determined using a novel automated measurement method. The colour intensity, which can be measured spectrophotometrically, is related to the total amount of oxidant molecules present in the sample. The assay is calibrated with hydrogen peroxide) and the results are expressed in terms of micromolar hydrogen peroxide equivalent per litre.
Device: Bispectral Index — Bispectral Index is a method for depth of anesthesia and assessment of sedation. The values of bispectral index decreases with the deepening of anesthesia. The values of 40-60 characterize the appropriate depth of anesthesia.
Other: Invasive arterial monitorization — Invasive arterial monitorization will be performed to right radial artery under local anesthesia to follow up hemodynamic changes and take the blood samples.

SUMMARY:
With the development of technology, the safety of anesthesia devices and the progression of monitoring techniques affect the anesthetic management. There are some disadvantages such as high cost of inhalation anesthetics and long postoperative recovery time. The effects of total intravenous anesthesia (TIVA), which has been used for many years and whose positive aspects are well known, on antioxidant system in high risk patients such as morbid obese should be investigated. The aim of this study was to compare the effects of desflurane anesthesia and total intravenous anesthesia (TIVA) on the antioxidant system in morbidly obese patients undergoing bariatric surgery.

DETAILED DESCRIPTION:
Obesity is a chronic disease that negatively affects the quality and duration of life. It is one of the most important health problem in the world and very common in Turkey. Morbid obesity operations have started to be performed frequently in our country with the effective results obtained with the continuation of weight loss after being widely applied in Europe and the United States. In our country, with the increase of obesity, laparoscopic bariatric is preferred especially with low complication rates.

Inhalation anesthesia is still a major source of chemical hazard in the hospital environment due to the widespread use in operating rooms. Factors affecting the presence of anesthetic gases in the environment; device leakage, ventilation, fresh gas flow and operation of the air wasting system. Long-term exposure to anesthetic gases is known to adversely affect the health of the workers in the operating room.

It has been shown that many anesthetic agents produce free radicals and alter serum antioxidant levels in patients. Antioxidant enzymes clean free radicals. Free radicals induced by various diseases can trigger oxidative stress and result in increased oxidative products. It was reported that particularly desflurane induced oxidative stress and increased oxidative products. At the same time, it was reported that desflurane triggered local and systemic oxidative stress in the experimental studies, but propofol had antioxidant properties.

With the development of technology, the safety of anesthesia devices and the progression of monitoring techniques affect the anesthetic management. There are some disadvantages such as high cost of inhalation anesthetics and long postoperative recovery time. The effects of total intravenous anesthesia (TIVA), which has been used for many years and whose positive aspects are well known, on antioxidant system in high risk patients such as morbid obese should be investigated. The aim of this study was to compare the effects of desflurane anesthesia and total intravenous anesthesia (TIVA) on the antioxidant system in morbidly obese patients undergoing bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology score I-III,
* 18-65 years,
* BMI> 40

Exclusion Criteria:

* American Society of Anesthesiology IV,
* Under 18 years,
* Over 65 years,
* Obstetric patients,
* Uncontrolled diabetes mellitus, cardiovascular and pulmonary disease,
* Cerebrovascular disease,
* Patients who refused informed consent forms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-07-21 (Actual)

PRIMARY OUTCOMES:
Total Antioxidant Status | Total Antioxidant Status 15 minutes before the anesthesia (preoperative period)
  Total Antioxidant Status values will be determined using a novel automated measurement method. The colour intensity, which can be measured spectrophotometrically, is related to the total amount of oxidant molecules present in the sample. The assay is calibrated with hydrogen peroxide) and the results are expressed in terms of micromolar hydrogen peroxide equivalent per litre.
Total Antioxidant Status | Total Antioxidant Status during the anesthesia (perioperative period, 60 minutes after the anesthesia induction)
  Total Antioxidant Status values will be determined using a novel automated measurement method. The colour intensity, which can be measured spectrophotometrically, is related to the total amount of oxidant molecules present in the sample. The assay is calibrated with hydrogen peroxide) and the results are expressed in terms of micromolar hydrogen peroxide equivalent per litre.
Total Antioxidant Status | Total Antioxidant Status after the anesthesia (postoperative period, 120 minutes after the surgery)
  Total Antioxidant Status values will be determined using a novel automated measurement method. The colour intensity, which can be measured spectrophotometrically, is related to the total amount of oxidant molecules present in the sample. The assay is calibrated with hydrogen peroxide) and the results are expressed in terms of micromolar hydrogen peroxide equivalent per litre.
Total Oxidant Status | 120 minutes
  Total Oxidant Status values will be determined using a novel automated measurement method. The colour intensity, which can be measured spectrophotometrically, is related to the total amount of oxidant molecules present in the sample. The assay is calibrated with hydrogen peroxide) and the results are expressed in terms of micromolar hydrogen peroxide equivalent per litre.
Total Oxidant Status | Total Oxidant Status during the anesthesia (perioperative period, 60 minutes after the anesthesia induction)
  Total Oxidant Status values will be determined using a novel automated measurement method. The colour intensity, which can be measured spectrophotometrically, is related to the total amount of oxidant molecules present in the sample. The assay is calibrated with hydrogen peroxide) and the results are expressed in terms of micromolar hydrogen peroxide equivalent per litre.
Total Oxidant Status | Total Oxidant Status after the anesthesia (postoperative period, 120 minutes after the surgery)
  Total Oxidant Status values will be determined using a novel automated measurement method. The colour intensity, which can be measured spectrophotometrically, is related to the total amount of oxidant molecules present in the sample. The assay is calibrated with hydrogen peroxide) and the results are expressed in terms of micromolar hydrogen peroxide equivalent per litre.

SECONDARY OUTCOMES:
Heart rate | From beginning of anesthesia (15 minutes before anesthesia) to end of anesthesia (15 minutes after anesthesia) up to nearly 5 hours]
  Heart rate (beat/min)
Mean Arterial Pressure | From beginning of anesthesia (15 minutes before anesthesia) to end of anesthesia (15 minutes after anesthesia) up to nearly 5 hours
  Mean Arterial Pressure (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Sedat Akbas, Asst. Prof., Principal Investigator — Inonu University Medical Faculty
Locations (1):
- Sedat Akbas, Malatya, Türkiye-Türkçe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han C, Ding W, Jiang W, Chen YU, Hang D, Gu D, Jiang G, Tan Y, Ge Z, Ma T. A comparison of the effects of midazolam, propofol and dexmedetomidine on the antioxidant system: A randomized trial. Exp Ther Med. 2015 Jun;9(6):2293-2298. doi: 10.3892/etm.2015.2410. Epub 2015 Apr 7. PMID 26136976

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT03814577/Prot_SAP_000.pdf